CLINICAL TRIAL: NCT00907101
Title: Evaluation of the Effectiveness of Epiduo® Gel (Adapalene 0.1% / Benzoyl Peroxide 2.5% Gel) in Reducing Antibiotic Sensitive and Resistant Strains of P Acnes
Brief Title: Evaluate Effectiveness of Epiduo® Gel in Reducing Antibiotic Sensitive & Resistant Strains of Propionibacterium (P)Acnes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: US10127
Record Dates: First submitted 2009-05-20; First posted 2009-05-22 (Estimated); Results first posted 2016-03-16 (Estimated); Last update posted 2022-08-01 (Actual); Status verified 2016-02

CONDITIONS: P Acnes Colonization
MeSH Terms: interventions — Adapalene; Benzoyl Peroxide; Gels

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Treatment (Experimental): Adapalene 0.1%/Benzoyl Peroxide 2.5% Gel (Epiduo® Gel)
  Other Names:
  Epiduo® Gel Apply once daily
  Interventions: Drug: Adapalene 0.1%/Benzoyl Peroxide 2.5% Gel (Epiduo® Gel)

INTERVENTIONS:
Drug: Adapalene 0.1%/Benzoyl Peroxide 2.5% Gel (Epiduo® Gel) — Apply once daily
  Other Names: Epiduo® Gel

SUMMARY:
The purpose of this study is to evaluate the effectiveness of Epiduo® Gel in reducing antibiotic sensitive and resistant strains of P acnes in vivo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male or female subjects 18 years of age and older, with no past or present history of any significant internal disease
* Subjects who:

  * show a high degree of fluorescence of the facial skin under a Wood's lamp, indicating the presence of P acnes
  * have Baseline P acnes count of > 10,000 per cm2 CFU of the facial skin (forehead)
  * have high level resistance to erythromycin, variable resistance to clindamycin, resistance to tetracycline and variable resistance to doxycycline and minocycline

Exclusion Criteria:

* Subjects who exhibit any skin disorders of an acute or chronic nature (e.g., psoriasis, eczema, etc)
* Subjects who have taken topical or systemic antibiotics within 4 weeks prior to baseline assessments
* Subjects who have used other medications which may influence skin surface P acnes levels
* Subjects who are unwilling to refrain from using toners, astringents or other drying agents on the face during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-06; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald W Gottschalk, MD, Study Director — Galderma R&D
Locations (1):
- Skin Study Center, Broomall, Pennsylvania, United States

REFERENCES:
- [Derived] Leyden JJ, Preston N, Osborn C, Gottschalk RW. In-vivo Effectiveness of Adapalene 0.1%/Benzoyl Peroxide 2.5% Gel on Antibiotic-sensitive and Resistant Propionibacterium acnes. J Clin Aesthet Dermatol. 2011 May;4(5):22-6. PMID 21607190

RESULTS

PARTICIPANT FLOW:
Groups:
- Epiduo® Gel: Adapalene 0.1%/Benzoyl Peroxide 2.5% Gel (Epiduo® Gel Applied Once Daily
Period: Overall Study
Arm/Group | Epiduo® Gel
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Epiduo® Gel
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.0 (12.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 29
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Skin Type [Number; unit: participants]
  Dry | 3
  Normal | 11
  Oily | 5
  Combination | 11
Fitzpatrick Skin Type [Number; unit: participants] — Investigator assessment based on the standard Fitzpatrick Skin Type Scale (I to VI).
  TYPE 1: Highly sensitive, always burns, never tans. TYP E 2: Very sun sensitive, burns easily, tans minimally. TYPE 3: Sun sensitive skin, sometimes burns, slowly tans to light brown. TYPE 4: Minimally sun sensitive, burns minimally, always tans to moderate brown.
  TYPE 5: Sun insensitive skin, rarely burns, tans well. TYPE 6: Sun insensitive, never burns, deeply pigmented.
  participants
    I | 0
    II | 3
    III | 12
    IV | 12
    V | 3
    VI | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Quantitative Bacteriology Measurements at Week 4
Description: Mean log10 values of P. acnes from swabbed skin samples Please note: Quantitative bacteriologic cultures were obtained from the facial skin (forehead) at screening, baseline, week 2 and week 4/early termination. Samples were obtained according to a modification of the technique of Williamson and Kligman. CFUs of P. acnes were counted at the dilution that contained between 10 and 100 CFUs. Total densities of P. acnes were calculated and reported as the average (of both plates) of the log10 CFUs per cm².
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: log10 CFU/cm2
Arm/Group | Epiduo® Gel
Number analyzed (Participants) | 30
log10 CFU/cm2 | -1.6 (0.78)

2. Secondary Outcome: Worst Post Baseline Tolerability Assessment - Erythema
Description: Please note: Tolerability assessments were recorded separately from adverse events. Tolerability changes which may have required a temporary or permanent interruption of the subject's participation in the study (at his/her request or at the investigator's discretion), or concomitant treatment, was to be recorded in the AE form of the CRF. An entry was to be made on the AE form for all AEs.
Time Frame: Week 4
Measure: Number; unit: participants
Arm/Group | Epiduo® Gel
Number analyzed (Participants) | 30
participants
  None | 30
  Mild | 0

3. Secondary Outcome: Worst Post Baseline Tolerability Assessment - Dryness
Description: as for outcome 2
Time Frame: Week 4
Measure: Number; unit: participants
Arm/Group | Epiduo® Gel
Number analyzed (Participants) | 30
participants
  None | 26
  Mild | 4

4. Secondary Outcome: Worst Post Baseline Tolerability Assessment - Scaling
Description: as for outcome 2
Time Frame: Week 4
Measure: Number; unit: participants
Arm/Group | Epiduo® Gel
Number analyzed (Participants) | 30
participants
  None | 29
  Mild | 1

5. Secondary Outcome: Worst Post Baseline Tolerability Assessment - Stinging/Burning
Description: as for outcome 2
Time Frame: Week 4
Measure: Number; unit: participants
Arm/Group | Epiduo® Gel
Number analyzed (Participants) | 30
participants
  None | 29
  Mild | 1

ADVERSE EVENTS:
Time Frame: Safety assessments were conducted for all subjects during each visit (baseline, week 2, week 4/early termination) after enrollment in the study
Description: No AEs were reported during the course of the study.
Arm/Group | Epiduo® Gel
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days